CLINICAL TRIAL: NCT00874523
Title: A Randomised, Open-label, Cross-over Study to Examine the Pharmacokinetics and Short-term Safety and Efficacy of Two Dosing Strategies of Raltegravir Plus Atazanavir in HIV-infected Patients
Brief Title: Raltegravir and Atazanavir Dosing Strategy Study
Acronym: SPARTA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kirby Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SPARTA
Record Dates: First submitted 2009-03-31; First posted 2009-04-02 (Estimated); Last update posted 2012-04-12 (Estimated); Status verified 2010-04

CONDITIONS: HIV Infection
Keywords: raltegravir; atazanavir; HIV infections; pharmacokinetics; antiretroviral agents; treatment experienced
MeSH Terms: conditions — HIV Infections | interventions — Atazanavir Sulfate; Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Active Comparator)
  Interventions: Drug: atazanavir plus raltegravir
- Arm B (Active Comparator)
  Interventions: Drug: atazanavir plus raltegravir

INTERVENTIONS:
Drug: atazanavir plus raltegravir — atazanavir 300 mg + raltegravir 400 mg twice daily for 4 weeks then atazanavir 300 mg + ritonavir 100 mg + raltegravir 800 mg once daily for 4 weeks
  Other Names: Reyataz; Isentress
  Arms: Arm A
Drug: atazanavir plus raltegravir — atazanavir 300 mg + ritonavir 100 mg + raltegravir 800 mg once daily for 4 weeks then atazanavir 300 mg + raltegravir 400 mg twice daily for 4 weeks
  Other Names: Reyataz; Isentress
  Arms: Arm B

SUMMARY:
To compare the steady-state pharmacokinetics and short-term efficacy and safety of two dosing strategies of raltegravir and atazanavir in virologically suppressed HIV-infected adults receiving atazanavir-containing combination antiretroviral therapy.

DETAILED DESCRIPTION:
Current HIV treatment guidelines recommend the construction of combination regimens comprising a minimum of three agents from at least two drug classes. There are problems with the current recommendations for although treatments are effective, their success is often limited by tolerability, adverse effects and the need to take many pills. Antiretroviral adherence remains vital and regimens should be simplified wherever possible to facilitate maximal adherence. The recent availability of the potent HIV integrase inhibitor, raltegravir, provides an opportunity to explore moves away from current regimen components. Evidence to support the use of novel regimens must be generated through adequately powered randomized clinical trials. However, before such trials can be undertaken, preliminary data to define the pharmacokinetics, safety and tolerability of these regimens are needed to minimize unnecessary risk for participants. This eight week study will investigate the steady-state pharmacokinetics, and short-term safety and efficacy of two dosing strategies (once and twice daily) of raltegravir plus atazanavir in treatment experienced HIV-infected adults.

ELIGIBILITY:
Inclusion Criteria:

* aged ≥ 18 years with laboratory evidence of HIV-1 infection
* currently receiving 3 or more unchanged antiretroviral agents including atazanavir (with or without ritonavir boosting) for at least 24 weeks prior to study entry
* plasma HIV RNA less than 50 copies/mL for at least 24 weeks prior to study entry
* provide written, informed consent.

Exclusion Criteria :

* prior clinical/virological failure on a PI-containing regimen
* no clinical history of primary HIV-1 protease mutations identified in local baseline genotypic analysis of HIV with interpretation using current IAS-USA Drug Resistance Mutations in HIV-1
* women: pregnant, breastfeeding, or not willing to use adequate contraception (including barrier contraception) if of child-bearing potential
* laboratory abnormalities at screening:

  * absolute neutrophil count (ANC) < 750 cells/mL
  * haemoglobin less than 8.5 g/dL
  * platelet count less than 50 000 cells/mL
  * AST, ALT > 5 times the upper limit of normal
  * serum bilirubin > 5 times the upper limit of normal
* chronic active hepatitis B infection defined by presence of serum viral hepatitis B surface antigen (HBsAg) or HBV DNA-positive
* any malabsorption syndrome likely to affect drug absorption
* concurrent therapy with human growth hormone or other immunomodulatory agents
* concomitant medication contraindicated for use with either atazanavir or raltegravir therapy
* any inter-current illness requiring hospitalisation
* current excessive alcohol or illicit substance use
* unlikely to be able to remain in follow-up for the protocol-defined period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2009-07; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
comparison of the mean steady-state atazanavir trough plasma concentrations for once (C24) and twice (C12) daily dosing strategies | 4 and 8 weeks

SECONDARY OUTCOMES:
comparison of mean steady-state raltegravir trough plasma concentrations for once (C24) and twice (C12) daily dosing | 4 and 8 weeks
comparison of steady-state pharmacokinetic profiles of once and twice-daily atazanavir | 4 and 8 weeks
comparison of the steady-state pharmacokinetic profiles of once and twice-daily raltegravir | 4 and 8 weeks
change from baseline in fasting lipid and glycaemic parameters | weeks 4 and 8 and overall
change from baseline in CD4+ T-lymphocyte count | weeks 4 and 8 and overall
change from baseline in HIV-RNA | weeks 4 and 8 and overall
all adverse events attributable to study treatment | week 8
all serious, grade 3 or 4 clinical adverse events, and any adverse event leading to premature cessation of study treatment | week 8

CONTACTS AND LOCATIONS:
Overall Officials: David A Cooper, MD DSc, Principal Investigator — Kirby Institute
Locations (2):
- Australia (2):
  - Holdsworth House Medical Practice, Sydney, New South Wales
  - St Vincent's Hospital, Sydney, New South Wales